CLINICAL TRIAL: NCT01717378
Title: Facilitating Enrollment Into UCSF Clinical Studies Via a Volunteer Research Participant Registry
Brief Title: UCSF Research Participant Registry
Status: Terminated | Type: Observational
Why Stopped: This is a voluntary registry formerly managed by a unit within CTSI that was disbanded in 2013. The registry has been dormant since that time.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 12-08393; UL1TR000004 (NIH)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Any Disease or Condition; Healthy
Keywords: Patient Recruitment; Research Subject Recruitment; Research Subject Selection; Selection of Subjects; Health Surveys; Health Questionnaires; Health Interviews

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Potential research participants: UCSF Registry represents a single recruitment pool of individuals who have consented to be contacted about future studies for which they may be eligible based on self-reported health information.

SUMMARY:
The UCSF Clinical and Translational Science Institute (CTSI) Consultation Service provides recruitment services and facilitates the enrollment of research participants into UCSF clinical studies. The Recruitment Services will be accessible to all researchers at UCSF and affiliated institutions and will address the common problems that investigators encounter in the recruitment process.

Recruitment Services considered and integrated Committee on Human Research (CHR) and HIPAA regulations for ensuring human subject rights, participant privacy, and data security into the recruitment workflow and data collection/extraction methods. Recruitment Services, therefore, requests approval to implement these processes systematically for all studies that have already obtained CHR approval to begin recruitment activities.

DETAILED DESCRIPTION:
The UCSF Research Participant Registry (http://registry.ucsf.edu) is a secure, standalone database that actively collects and stores data from willing volunteers who visit its website. The UCSF Registry is a cornerstone of the UCSF Recruitment Service (RS). Both the Registry and the RS are among several initiatives implemented by the UCSF Clinical & Translational Science Institute.

The chief purpose of the RS is to facilitate the enrollment of research participants into UCSF clinical studies. The primary function of the Registry is to expand the pool of potential clinical research volunteers. The Registry stores self-reported identifiable health information in a searchable database that is compliant with the privacy requirements of the Health Insurance Portability and Accountability Act (HIPAA). This information is then used by the RS for the future identification and recruitment of potentially eligible participants for specific UCSF studies.

Registry participants whose data matches the major eligibility criteria for a specific study will be sent recruitment materials about the study. Contact information for the investigator or RS staff will also be included in the e-mailing. Participants are then free to choose whether to respond or ignore the study recruitment information.

ELIGIBILITY:
INCLUSION CRITERIA

* Adults age 18 years or older
* Minors/children with consent from parent or guardian (Parents or guardians must provide their own contact information and then complete the questionnaire using the child's health information.)

EXCLUSION CRITERIA

* Failure to provide consent
* Minors/children without consent of parent or guardian

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General public. Anyone may join the UCSF Registry, but adult & pediatric residents of the San Francisco Bay Area are targeted because of their proximity to UCSF research clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1541 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Increased screening & enrollment for UCSF clinical studies | 4 years
  By broadening the pool of potential volunteers, the Registry is expected to increase the number of screened & enrolled participants in UCSF studies.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah G Grady, MD, MPH,FACP, Principal Investigator — Clinical & Translational Science Institute, University of California San Francisco
Locations (1):
- Clinical & Translational Science Institute, University of California San Francisco, San Francisco, California, United States

REFERENCES:
- See also: UCSF Research Participant Registry — http://registry.ucsf.edu